CLINICAL TRIAL: NCT01433614
Title: Treatment With the Combination of Epirubicin and Paclitaxel Alone or Together With Capecitabine as First Line Treatment in Metastatic Breast Cancer. A Multicenter, Randomized Phase III Study
Brief Title: Epirubicin and Paclitaxel, Alone or Together With Capecitabine as First Line Treatment in Metastatic Breast Cancer
Acronym: TEX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thomas Hatschek (Other)
Responsible Party: Sponsor-Investigator, Thomas Hatschek, MD, PhD, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEX trial
Record Dates: First submitted 2011-09-01; First posted 2011-09-14 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Epirubicin; Paclitaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epirubicin + paclitaxel (Taxol) (Active Comparator): Epirubicin 75mg/m2 i.v., paclitaxel 175 mg/m2 i.v. on day 1 every 21 days.
  Interventions: Drug: Epirubicin; Drug: Paclitaxel
- Paclitaxel + epirubicin + capecitabine (Active Comparator): Paclitaxel 155 mg/m2 i.v., epirubicin 75 mg/m2 i.v day 1, capecitabine 1650 mg/m2 p.o. on days 1-14 every 21 days.
  Interventions: Drug: Epirubicin; Drug: Paclitaxel; Drug: Capecitabine

INTERVENTIONS:
Drug: Epirubicin — 75 mg/m2 i.v. every 3 weeks, both study arms
Drug: Paclitaxel — 175 mg/m2 i.v., every 3 weeks study arm A 155 mg/m2 i.v., every 3 weeks study arm B
  Other Names: Taxol
Drug: Capecitabine — 1650 mg/m2 p.o. days 1-14 every 3 weeks study arm B
  Other Names: Xeloda
  Arms: Paclitaxel + epirubicin + capecitabine

SUMMARY:
Anthracycline-taxane regimens are effective means of postponing progression in metastatic breast cancer. It is yet unclear whether addition of capecitabine to this combination improves the treatment outcome.

Patients with advanced breast cancer are randomized to first-line chemotherapy with a combination of epirubicin (Farmorubicin®) and paclitaxel (Taxol®) alone (ET) or in combination with capecitabine (Xeloda®, TEX). Starting doses for ET are epirubicin 75 mg/m2 plus paclitaxel 175 mg/m2, and for TEX epirubicin 75mg/m2, paclitaxel 155 mg/m2, and capecitabine 825 mg/m2 BID for 14 days. Subsequently, doses are tailored related to side effects.

Primary endpoint is progression-free survival (PFS); secondary endpoints are overall survival (OS), time to treatment failure (TTF), objective response (OR), safety and quality of life (QoL).

ELIGIBILITY:
Inclusion Criteria:

* Morphologically proven breast carcinoma
* Written patient consent must be obtained
* Measurable disease (i.e. at least one lesion that can be accurately measured in at least one dimension as ≥20 mm by conventional techniques, or as ≥10 mm by spiral CT scan) as defined in section 8.
* Lytic and blastic bone metastases as only site of recurrence are allowed
* Age 18 years or older
* ECOG performance status 0-2
* Life expectancy of at least three months
* Adequate cardiac functions
* Adequate hematological, renal and hepatic functions
* Patient must be accessible for treatment and follow-up.

Exclusion Criteria:

* Treatment-free interval less than one year, if previous adjuvant, neoadjuvant or after radically treated locoregional recurrence given regimen contained anthracycline, taxane or capecitabine. This limitation does not apply for regimens containing other than the drugs mentioned
* During adjuvant treatment obtained cumulative doses exceeding 375 mg/m2 for doxorubicin, or 550 mg/m2 for epirubicin, abnormal ECG or reduced cardiac function measured by left ventricular ejection fraction (LVEF).
* Indication for the use of trastuzumab (Herceptin) as first-line treatment in patients with tumor overexpressing c-erbB2.
* Any previous chemotherapy for metastatic disease, except for radically treated locoregional relapse
* Neoplasm other than breast carcinoma, except for non-melanoma skin cancer or curatively treated carcinoma in situ of the cervix, diagnosed during the past five years
* Pregnancy or lactation
* Known brain metastases
* History of atrial or ventricular arrhythmias and/or congestive heart failure, even if medically controlled. History of clinical and electrocardiographically documented myocardial infarction
* Preexisting motor or sensory neuropathy ≥ grade 2 according to NCI CTC 2.0 criteria (severe paresthesia and/or mild weakness, or worse)
* Severe hepatic or renal impairment (for capecitabine: calculated creatinine clearance below 30 ml/min; for calculation, see p. 5.1.4) not allowing for adequate use of the proposed regimens
* History of known dihydropyrimidine dehydrogenase (DPD) deficiency (severe reaction on previous treatment with fluorouracil, e.g experience of mucositis, hand-foot syndrome, or diarrhea)
* Active infection or other serious underlying medical condition which would impair the ability of the patient to receive protocol treatment, including prior allergic reactions to drugs containing cremophor, such as teniposide, cyclosporin or vitamin K
* Dementia or significantly altered mental status that would prohibit the understanding and giving of informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2002-12; Primary Completion 2006-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Time to progression | From date of randomisation until date of first radiolocically documented progression or death from any cause, whichever comes first up to 78 months
  Time to progression comparing treatment with ET vs. TEX in patients with advanced breast cancer. Evaluation every 9 weeks during treatment until progression as long as study treatment was given, and every 12 weeks until date of progression, if treatment was disrupted for any other reason. Patients in the state of persistent complete response after primary completion date were reported only upon date of progression or death up to 78 months

SECONDARY OUTCOMES:
Time to treatment failure | From date of randomization until date of treatment disruption for any reason up to 78 months
  Time on treatment irrespective of reason for disruption (toxicity, patients wish)
Response rate | Every 9 weeks during treatment
Overall survival | Time from randomisation until date of death up to 78 months
  Date and cause of death reported yearly during the ongoing trial, up to 78 months after primary completion date only on the occasion of death
Number of participants with adverse events | Continuously during treatment and until 2 months after termination
  All side effects which appear during treatment are reported and graded according CTC v.2.
Quality of life | Baseline, 2, 4, 6 and 9 months
  Measured at five points during nine months from randomization.
Tumor biological data related to treatment | Within two weeks before start of treatment
  Fine needle aspirates from metastases

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hatschek, PhD, Principal Investigator — Karolinska University Hospital
Locations (9):
- Sweden (9):
  - Sahlgrenska University Hospital, Gothenburg
  - Helsingborg Gen. Hospital, Helsingborg
  - Kalmar Central Hospital, Kalmar
  - Karlstad Gen. Hospital, Karlstad
  - Linköping University Hospital, Linköping
  - Lund University Hospital, Lund
  - Malmö General University Hospital, Malmo
  - Sundsvall Gen. Hospital, Sundsvall
  - Norrland University Hospital, Umeå

REFERENCES:
- [Result] Svensson H, Brandberg Y, Einbeigi Z, Hatschek T, Ahlberg K. Psychological reactions to progression of metastatic breast cancer--an interview study. Cancer Nurs. 2009 Jan-Feb;32(1):55-63. doi: 10.1097/01.NCC.0000343374.09270.ff. PMID 19104202
- [Result] Svensson H, Einbeigi Z, Johansson H, Hatschek T, Brandberg Y. Quality of life in women with metastatic breast cancer during 9 months after randomization in the TEX trial (epirubicin and paclitaxel w/o capecitabine). Breast Cancer Res Treat. 2010 Oct;123(3):785-93. doi: 10.1007/s10549-010-1084-8. Epub 2010 Aug 3. PMID 20680680
- [Result] Svensson H, Hatschek T, Johansson H, Einbeigi Z, Brandberg Y. Health-related quality of life as prognostic factor for response, progression-free survival, and survival in women with metastatic breast cancer. Med Oncol. 2012 Jun;29(2):432-8. doi: 10.1007/s12032-011-9844-9. Epub 2011 Feb 6. PMID 21298494
- [Result] Hatschek T, Carlsson L, Einbeigi Z, Lidbrink E, Linderholm B, Lindh B, Loman N, Malmberg M, Rotstein S, Soderberg M, Sundquist M, Walz TM, Hellstrom M, Svensson H, Astrom G, Brandberg Y, Carstensen J, Ferno M, Bergh J. Individually tailored treatment with epirubicin and paclitaxel with or without capecitabine as first-line chemotherapy in metastatic breast cancer: a randomized multicenter trial. Breast Cancer Res Treat. 2012 Feb;131(3):939-47. doi: 10.1007/s10549-011-1880-9. Epub 2011 Nov 18. PMID 22094937
- [Result] Suzuki C, Blomqvist L, Hatschek T, Carlsson L, Einbeigi Z, Linderholm B, Lindh B, Loman N, Malmberg M, Rotstein S, Soderberg M, Sundqvist M, Walz TM, Astrom G, Fujii H, Jacobsson H, Glimelius B. Impact of the first tumor response at eight weeks on overall survival in metastatic breast cancer patients treated with first-line combination chemotherapy. Med Oncol. 2013 Mar;30(1):415. doi: 10.1007/s12032-012-0415-5. Epub 2013 Jan 16. PMID 23322522
- [Result] Bjohle J, Bergqvist J, Gronowitz JS, Johansson H, Carlsson L, Einbeigi Z, Linderholm B, Loman N, Malmberg M, Soderberg M, Sundquist M, Walz TM, Ferno M, Bergh J, Hatschek T. Serum thymidine kinase activity compared with CA 15-3 in locally advanced and metastatic breast cancer within a randomized trial. Breast Cancer Res Treat. 2013 Jun;139(3):751-8. doi: 10.1007/s10549-013-2579-x. Epub 2013 Jun 5. PMID 23736998
- [Result] Tobin NP, Harrell JC, Lovrot J, Egyhazi Brage S, Frostvik Stolt M, Carlsson L, Einbeigi Z, Linderholm B, Loman N, Malmberg M, Walz T, Ferno M, Perou CM, Bergh J, Hatschek T, Lindstrom LS; TEX Trialists Group. Molecular subtype and tumor characteristics of breast cancer metastases as assessed by gene expression significantly influence patient post-relapse survival. Ann Oncol. 2015 Jan;26(1):81-88. doi: 10.1093/annonc/mdu498. Epub 2014 Oct 31. PMID 25361981
- [Result] Kimbung S, Kovacs A, Bendahl PO, Malmstrom P, Ferno M, Hatschek T, Hedenfalk I. Claudin-2 is an independent negative prognostic factor in breast cancer and specifically predicts early liver recurrences. Mol Oncol. 2014 Feb;8(1):119-28. doi: 10.1016/j.molonc.2013.10.002. Epub 2013 Oct 14. PMID 24287398
- [Result] Kimbung S, Johansson I, Danielsson A, Veerla S, Egyhazi Brage S, Frostvik Stolt M, Skoog L, Carlsson L, Einbeigi Z, Lidbrink E, Linderholm B, Loman N, Malmstrom PO, Soderberg M, Walz TM, Ferno M, Hatschek T, Hedenfalk I; TEX study group. Transcriptional Profiling of Breast Cancer Metastases Identifies Liver Metastasis-Selective Genes Associated with Adverse Outcome in Luminal A Primary Breast Cancer. Clin Cancer Res. 2016 Jan 1;22(1):146-57. doi: 10.1158/1078-0432.CCR-15-0487. Epub 2015 Aug 14. PMID 26276891
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241